CLINICAL TRIAL: NCT01909908
Title: Treatment of Chronic Wounds Using Extracellular Matrix-Based Devices and the Patient's Own Blood Components
Brief Title: ECM and Blood Components for Wound Healing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-014
Record Dates: First submitted 2013-07-25; First posted 2013-07-29 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Ulcer; Venous Ulcer; Foot Ulcer, Diabetic
Keywords: Wounds and injuries; Ulcer; Diabetic angiopathies; Diabetic foot; Venous insufficiency; Extracellular matrix
MeSH Terms: conditions — Ulcer; Varicose Ulcer; Diabetic Foot; Wounds and Injuries; Diabetic Angiopathies; Venous Insufficiency

ARMS (3):
- ECM in Saline (Experimental)
  Interventions: Device: ECM
- Blood Products (Active Comparator)
  Interventions: Biological: Blood Products
- ECM in Blood Products (Experimental)
  Interventions: Device: ECM in Blood Products

INTERVENTIONS:
Device: ECM — ECM in saline applied to wound
  Arms: ECM in Saline
Biological: Blood Products — Autologous blood product applied to wound, with saline cleanse on alternating weeks
  Arms: Blood Products
Device: ECM in Blood Products — Alternating treatments of ECM in saline and ECM in autologous blood products, applied to wound
  Arms: ECM in Blood Products

SUMMARY:
The Extracellular Matrix (ECM) and Blood Components for Wound Healing feasibility study is a clinical trial approved by Health Canada to study the safety of extracellular matrix (ECM) and autologous blood products in wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or Type 2 diabetes, and/or venous insufficiency to the affected leg
* Ulcer has been present between 12 and 52 weeks
* Ulcer is less than 40 cm2 in area

Exclusion Criteria:

* Less than 18 years of age
* Pregnant or planning to become pregnant during the study period
* Simultaneously participating in another investigational drug or device study
* Unable or unwilling to comply with the weekly study follow-up schedule or off-loading regimen
* Patient or legal representative refuses to sign the EC-approved informed consent form
* Known allergy to pig or porcine products
* Additional criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-02; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Embil, MD, FRCPC, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada